CLINICAL TRIAL: NCT06616675
Title: Darifenacin Versus Parasacral Transcutaneous Electric Nerve Stimulation for Overactive Bladder Syndrome in Patients Infected With Human T-Lymphotropic Virus 1 - Randomized Open Clinical Trial
Brief Title: Darifenacin x Parasacral Transcutaneous Electric Nerve Stimulation for OAB in Patients Infected With Human T-Lymphotropic Virus 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Responsible Party: Principal Investigator, Tatiane Souza Soares de Oliveira, Physiotherapist, Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 59171022.9.0000.0049
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: HTLV-1; Overactive Bladder Syndrome
Keywords: Electrical stimulation; Overactive bladder; HLTV-1; darifenacin
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — darifenacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Darifenacin Group (Active Comparator): Anticholinergic treatment for OAB
  Interventions: Drug: Darifenacin
- PTENS Group (Experimental): Neuromodulation using transcutaneous electrical sacral nerves stimulation
  Interventions: Device: Neuromodulation - Sacral nerve stimulation

INTERVENTIONS:
Drug: Darifenacin — Anticholinergic drug therapy for OAB treatment - Darifenacin, 15mg/day
  Arms: Darifenacin Group
Device: Neuromodulation - Sacral nerve stimulation — Neurodyn Portable TENS FES neuromuscular stimulation device in an outpatient clinic. Two self-adhesive electrodes (5x9cm) were used, positioned one in each gluteal region, below the iliac spine to apply low-frequency biphasic current with 10 Hz. Pulse duration of 0.5 milliseconds was applied for 40 minutes with continuous stimulation, 3 times a week, for 20 sessions.
  Arms: PTENS Group

SUMMARY:
In this study the investigators compare the parasacral transcutaneous electric nerve stimulation (PTENS) treatment with Darifenacin to improve OAB symptoms in patients infected with HTLV-1.

DETAILED DESCRIPTION:
Subjects presenting OAB according to ICS, associated with the HTLV-1 infection were invited by the investigators to participate in the study according inclusion criteria . Participants who accepted were randomly allocated to two groups (G1 and G2) by the free randomization website. Group 1 was treated with Darifenacin, and group 2 with the PTENS protocol.

Drug Treatment Protocol:

The anticholinergic Fenazic (Adium) was used in a single dose of 15mg/day for 2 months.

PTENS Protocol:

The treatment consisted of PTENS with the Neurodyn Portable TENS FES(21) neuromuscular stimulation device in an outpatient clinic. Two self-adhesive electrodes (5x9cm) were used, positioned one in each gluteal region, below the iliac spine to apply low-frequency biphasic current with 10 Hz. Pulse duration of 0.5 milliseconds was applied for 40 minutes with continuous stimulation, 3 times a week, for 20 sessions.

ELIGIBILITY:
Inclusion Criteria:

* HTLV-1 infection
* Overactive bladder symptom
* 18 years of age or older

Exclusion Criteria:

* HTLV-1 infected subjects with HAM
* Stroke
* Parkinson
* HIV infection
* Prostatic hyperplasia
* Pacemaker use
* Genitourinary tract infection
* Glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Overactive Bladder Symptom Score | 2 months or 20 sessions
  Whether higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Ambulatório de HTLV-1 - Com HUPES, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu Y, Xu G, Geng J. Efficacy of Transcutaneous Electrical Nerve Stimulation in the Management of Neurogenic Overactive Bladder: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2022 Jan 1;101(1):2-10. doi: 10.1097/PHM.0000000000001836. PMID 34225282
- [Result] Slovak M, Chapple CR, Barker AT. Non-invasive transcutaneous electrical stimulation in the treatment of overactive bladder. Asian J Urol. 2015 Apr;2(2):92-101. doi: 10.1016/j.ajur.2015.04.013. Epub 2015 Apr 16. PMID 29264126
- [Result] Andrade RC, Neto JA, Andrade L, Oliveira TS, Santos DN, Oliveira CJ, Prado MJ, Carvalho EM. Effects of Physiotherapy in the Treatment of Neurogenic Bladder in Patients Infected With Human T-Lymphotropic Virus 1. Urology. 2016 Mar;89:33-8. doi: 10.1016/j.urology.2015.09.036. Epub 2015 Dec 24. PMID 26724409